CLINICAL TRIAL: NCT03706027
Title: Three- Versus Five-Fraction Regimens of Stereotactic Body Radiotherapy for Peripheral Early-Stage Non-Small-Cell Lung Cancer: A Prospective Randomized Phase II Study
Brief Title: Study Comparing Two Different Schedules of Radiation for Early-stage Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Deepinder P Singh, MD, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72835
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stereotactic body radiotherapy- 3 fractions (Active Comparator)
  Interventions: Device: radiation therapy-3 fractions
- Stereotactic body radiotherapy- 5 fractions (Active Comparator)
  Interventions: Device: Radiation therapy-5 fractions

INTERVENTIONS:
Device: radiation therapy-3 fractions — Radiation therapy given in a 3 fraction schedule (over 3 days). Total dose is 54 Grays.
  Arms: Stereotactic body radiotherapy- 3 fractions
Device: Radiation therapy-5 fractions — Radiation therapy given in 5 fractions (over 5 days). Total dose is 60 Grays.
  Arms: Stereotactic body radiotherapy- 5 fractions

SUMMARY:
This study's goal is to find out if the kind of side effects people experience from radiation is different depending on the schedule of their radiation treatment. Patients will be randomly assigned to either the 3 Fraction or 5 Fraction schedule of radiation. After patients complete radiation treatment, they will follow up with their radiation oncologist.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of non-small cell cancer will not be required as primary goal of this phase II trial is to look at toxicity. However, all primary non-small cell lung cancers otherwise of following types are eligible: squamous cell carcinoma, adenocarcinoma, large cell carcinoma, bronchioalveolar cell carcinoma, or non-small cell carcinoma not otherwise specified.
* Eligible patients must have appropriate staging studies identifying them as specific subsets of AJCC stage I or II based on only one of the following combinations of TNM staging:
* T1, N0, M0
* T2 (≤ 5 cm), N0, M0
* Patients with hilar or mediastinal lymph nodes ≤ 1cm and no abnormal hilar or mediastinal uptake on PET will be considered N0. Patients with > 1 cm hilar or mediastinal lymph nodes on CT or abnormal PET (including suspicious but non-diagnostic uptake) may still be eligible if directed tissue biopsy of all abnormally identified areas are negative for cancer. All patients with suspicious nodes will be evaluated for mediastinal and hilar staging with bronchoscopy and (if amenable) bronchoscopic biopsy (preferably navigational biopsy and/or endobronchial US guided biopsy).
* Zubrod performance status 0-2 within 4 weeks of study entry.
* Women of childbearing potential and male participants must use an effective contraceptive method.
* Evaluations required at time of study entry:
* History & Physical by a radiation oncologist within 4 weeks of study entry;
* Vitals within 4 weeks of study entry;
* Evaluation by a thoracic surgeon (either via clinical examination and/or input at multidisciplinary tumor board) prior to study entry;
* PFTs: Routine spirometry, lung volumes, diffusion capacity, and arterial blood gases within 8 weeks prior to study entry;
* CT Chest within 6 weeks of study entry (preferably with intravenous contrast, unless medically contraindicated) - to include the entirety of both lungs, the mediastinum, liver, and adrenal glands; primary tumor dimension will be measured on this CT;
* Whole body positron emission tomography (PET) scan using FDG with adequate visualization of the primary tumor and draining lymph node basins in the hilar and mediastinal regions within 6 weeks prior to study entry.
* Informed consent signed by the subject and a member of the study team.

Exclusion Criteria:

* Patients with central tumors. Specifically; central location implies a tumor inside the zone of the proximal bronchial tree defined as a volume 2 cm in all directions around the proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus, right and left lower lobe bronchi
* Evidence of regional or distant metastases after appropriate staging studies.
* Synchronous primary NSCLC.
* Those with prior malignancy in the past 2 years other than non-melanomatous skin cancer or in situ cancer or thyroid cancer.
* Previous lung or mediastinal radiotherapy.
* Plans for the patient to receive concomitant antineoplastic therapy (including standard fractionated radiotherapy, chemotherapy, biological therapy, vaccine therapy, and surgery) while on this protocol.
* Patients with active systemic, pulmonary or pericardial infection.
* Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
frequency of grade 3 treatment related toxicities or higher | 1 year
  Toxicities will be assessed using the National Cancer Institute common toxicities criteria version 4.0. The rates of grade 3 or higher adverse events at 1 year will be calculated as the proportion of patients who have any adverse event of interest by the end of year 1 among the total analyzable patients in each arm.

SECONDARY OUTCOMES:
mean survival time of patients with overall survival | 3 years
  The failure event for overall survival is a death due to any cause. Survival time is measured from the date of randomization to the date of death or last follow up.
proportion of patients with disease-free survival | 3 years
  The failure event for disease-free survival is defined as death due to any cause, local failure, marginal failure, involved node failure, regional failure, distant metastasis, or second primary.
proportions of patients with primary tumor control | 3 years
  Marginal failures will be considered events for primary tumor failure. The primary tumor control rate at 1 year will be calculated as the number of patients who do not have a local progression event by the total number of analyzable patients in each arm at 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No